CLINICAL TRIAL: NCT03038269
Title: Transcranial Direct Current Stimulation and Robotic Training in Adults With Cerebral Palsy
Brief Title: tDCS and Robotic Training in Adults With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Principal Investigator, Kathleen Friel, Director, Clinical Laboratory for Early Brain Injury Recovery, Burke Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BRC 467
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy; Hemiplegia
Keywords: Robotics; Upper Extremity
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham tDCS (Sham Comparator): Participant will receive a placebo-type stimulation followed by upper extremity robotic training.
  Interventions: Behavioral: Upper Extremity Robotics, tDCS
- Active tDCS (Active Comparator): Participant will receive active transcranial direct current stimulation followed by upper extremity robotic training.
  Interventions: Behavioral: Upper Extremity Robotics, tDCS

INTERVENTIONS:
Behavioral: Upper Extremity Robotics, tDCS — Participant will receive 20 minutes of non-invasive brain stimulation followed by one hour of shoulder/wrist robotic training.

SUMMARY:
The purpose of this study is to improve arm function in adults with hemiplegic cerebral palsy. Participants will receive transcranial direct current stimulation (or sham) in combination with upper extremity robotic therapy.

DETAILED DESCRIPTION:
Therapy consists of 20 minutes of non-invasive, low-level brain stimulation (transcranial direct current stimulation, tDCS), followed by one hour of shoulder/wrist robotic training. Participants will be enrolled in therapy 3 times per week for 12 weeks (or 36 sessions). Before and after therapy, participants will receive and assessment of their arm function, as well as an assessment of their brain activity, using electroencephalography (EEG) and transcranial magnetic stimulation (TMS).

ELIGIBILITY:
Inclusion Criteria:

* Participant willing and able to provide informed consent
* Diagnosis of hemiplegic Cerebral Palsy
* Joint mobility: wrist extention (20 degrees), metacarophalangeal and proximal interphalangeal joints (10 degrees)

Exclusion Criteria:

* Cognitive deficits that impede understanding of study protocol
* Current medical illness unrelated to CP
* Visual problems (uncorrected by glasses/contact lenses)
* High motor ability in affected arm
* Severe spasticity
* Lack of asymmetry in hand function
* Orthopedic surgery in affected arm within 2 years
* Dorsal root rhizotomy
* Botulinum toxin therapy in either upper extremity during last 2 months, or planned during study period
* Currently receiving intrathecal baclofen
* Seizure beyond age 2, use of anti-seizure medication, history of epilepsy (in self or first degree relatives), brain surgery, cranial metal implants, structural brain lesion, deices that may be affected by TMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* True positive response on the Transcranial Magnetic Stimulation Safety Screen
* Current use of medications known to lower the seizure threshold
* Previous episode of neurocardiogenic snycopy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-12; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Motor Recovery | 1 Week
  Evaluates and measures recovery

SECONDARY OUTCOMES:
Wolf Motor Function Test | 1 Week
  Quantifies upper extremity motor ability through timed and functional tasks
Box and Blocks Test | 1 Week
  Measures unilateral gross motor dexterity.

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Friel KM, Lee P, Soles LV, Smorenburg ARP, Kuo HC, Gupta D, Edwards DJ. Combined transcranial direct current stimulation and robotic upper limb therapy improves upper limb function in an adult with cerebral palsy. NeuroRehabilitation. 2017;41(1):41-50. doi: 10.3233/NRE-171455. PMID 28505986